CLINICAL TRIAL: NCT06465654
Title: OXYWILD - Automated Oxygen Titration With O2matic During Walking in Patients With Fibrotic Interstitial Lung Diseases (F-ILD): A Randomized Study
Brief Title: Automated Oxygen Titration During Walking in Patients With Lung Fibrosis (OXYWILD)
Acronym: OXYWILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janne Hastrup Jensen (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor-Investigator, Janne Hastrup Jensen, Physiotherapist, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UAarhus_OXYWILD
Record Dates: First submitted 2024-05-27; First posted 2024-06-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fibrosis Lung; Respiratory Therapy
Keywords: Automated oxygen titration; Fibrotic interstitial lung disease; Walking test
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: In random order the participants will conduct the endurance shuttle walk test with either fixed dose oxygen treatment or automated oxygen titration treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant will wear a high flow nasal canula for oxygen treatment during both endurance shuttle walk tests, which will mask the mode of oxygen delivery and dose for both the participant and the assessor (investigator). A health care professional not involved in the data collection or outcome assessment will set up the equipment before each test to secure masking of the O2matic device and oxygen delivery mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endurance shuttle walk test with fixed dose oxygen treatment (Active Comparator): The participant will conduct an endurance shuttle walk test with a fixed oxygen dose of 4 liters/minute delivered by the O2matic.
  Interventions: Other: Fixed dose oxygen treatment
- Endurance shuttle walk test with automated variable dose oxygen treatment (Experimental): The participant will conduct an endurance shuttle walk test with closed loop oxygen titration using O2matic to deliver a variable oxygen dosage set at an oxygen saturation target of 90 to 94 percent and an oxygen flow of 4 - 15 liters/minute.
  Interventions: Other: Automated variable dose oxygen treatment

INTERVENTIONS:
Other: Automated variable dose oxygen treatment — The participant will receive closed loop oxygen titration during a walking test based on oxygen saturation measurements every second measured by a pulse oximeter connected to the O2matic. The participant will every minute during the walking test rate sensation of dyspnea on the BorgCR10 scale.
  Other Names: Closed loop oxygen titration with O2matic
  Arms: Endurance shuttle walk test with automated variable dose oxygen treatment
Other: Fixed dose oxygen treatment — The participant will receive a fixed oxygen dose during a walking test. The participant will every minute during the walking test rate sensation of dyspnea on the BorgCR10 scale.
  Arms: Endurance shuttle walk test with fixed dose oxygen treatment

SUMMARY:
Fibrotic lung disease is a group of severe scarring lung diseases with a dismal prognosis, often leading to respiratory failure and need for oxygen treatment. The symptom burden is often extremely high with dyspnea at rest and increasing dyspnea with exertion. Patients will often need more oxygen during activity thus repeatedly adjustments of oxygen flow rates are required to target an acceptable saturation at rest and during activities. This is impractical and can lead to an undesirable focus on oxygen levels as well as reduced use of the oxygen treatment in everyday life.

There is an urgent need for oxygen equipment that is easy to use to help patients live a life with fever symptom-related restrictions. Closed Loop Oxygen Titration (CLOT) is a new type of optimized oxygen treatment, which automatically adjusts the oxygen flow rate to the exact amount needed for the patient. The CLOT has already been tested and found useful in patients with other lung diseases, however it has not yet been tested in an isolated group of patients with fibrotic lung disease.

The goal of this clinical trial is therefore to study if automatically adjusted oxygen delivery can be useful for patients with fibrotic lung disease who needs oxygen treatment during activity.

The main questions aimed to be answered are: Will participants experience less breathlessness during walking, when the oxygen supply is individually adjusted to maintain an acceptable level of oxygen saturation?

Our hypotheses are that automatically adjusted oxygen dose during walking will results in less breathlessness compared to the usual fixed dose of oxygen. Furthermore, that participants will walk longer and maintain a better oxygen saturation during a walking test when offered automatically adjusted oxygen dose.

Participants will perform two walking tests with both automatically adjusted and fixed dose oxygen in random order, and the difference in sensation of breathlessness will be compared between the two tests.

DETAILED DESCRIPTION:
Recruitment of participants

Participants with fibrotic lung disease will be recruited by a pulmonary specialist from the Centre for Rare Lung Diseases, Department of Respiratory Diseases and Allergy, Aarhus University Hospital during a routine outpatient visit. If exertional oxygen desaturation is suspected or has been documented by a six-minute walking test the investigator, a pulmonary specialist will inform the patient about the study and ask for study participation.

The patient will be asked to sign the informed consent. The information given to the patient specifies that the informed consent gives access for study personnel to access the medical record for relevant information necessary to complete the study. The written informed consent form will be signed and personally dated by the subject and the person conducting the informed consent conversation.

Ethical considerations

No risk for the patients is considered to be related to participation in the study. The walking tests are conducted by an experienced physiotherapist with solid knowledge about patients with fibrotic lung disease and when to terminate walking tests due to clinical symptoms. Furthermore, patients are enquired to stop the test if they experience discomfort. Walking tests with or without oxygen supply is a part of standard clinical practice for patients with fibrotic lung disease at the Centre of Rare Lung Diseases and the O2matic has been approved for clinical use.

Patients can benefit individually by gaining knowledge about their oxygen need at exercise, and as a group contribute to increased knowledge about the effect of automated oxygen treatment on dyspnea during exercise and on exercise endurance. International guidelines have restricted recommendations for ambulatory oxygen therapy due to limited evidence. This study may contribute to stronger recommendations for the prescription of ambulatory oxygen therapy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of fibrotic interstitial lung disease
* Desaturation during a recent (6 months) 6-minute walk test below 88% on atmospheric air or during an incremental shuttle walking test
* Able to walk at least 50 meters
* Self-reported stable respiratory symptoms in the previous 2 weeks
* Age ≥ 18 years
* Cognitively able to understand and participate in the study
* Written informed consent

Exclusion Criteria:

* Long term oxygen treatment
* A pulmonary or cardiac condition other than fibrotic interstitial lung disease limiting exercise performance
* Unstable heart condition or symptomatic stenotic valve disease
* Any physical condition limiting exercise performance.
* Smoking the previous 24 hours
* Pregnancy
* Anaemia, haemoglobin < 7.3 mmol/l (women) or < 8.3 mmol/l (men)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Borg dyspnea score | At baseline and through completion (one day)
  Primary outcome is the difference in Borg dyspnea score at isotime between the two endurance shuttle walk test (fixed dose oxygen compared to automated variable dose oxygen). The dyspnea score is rated every minute with the Borg Category-Ratio (CR)10 scale, where 0 is "no dyspnea at all" and 10 is "maximum dyspnea ever experienced".

SECONDARY OUTCOMES:
Walking distance | At baseline and through completion (one day)
  Difference in walking distance in meters between groups in Endurance shuttle walking test
Walking time | At baseline and through completion (one day)
  Difference in walking time in seconds between groups in Endurance shuttle walking test
Oxygen flow rate | At baseline and through completion (one day)
  Difference in average oxygen flow rate (liter/minute) between groups in Endurance shuttle walking test.
Oxygen saturation levels | At baseline and through completion (one day)
  Difference in time spent in seconds within acceptable oxygen saturation interval (oxygen saturation 90 - 94 percentage and time spent with moderate hypoxemia (oxygen saturation below 88 percentage) and severe hypoxemia (Oxygen saturation below 85 percentage) with moderate hypoxemia (oxygen saturation below 88 percentage) and severe hypoxemia (oxygen saturation below 85 percentage.
Hypoxemia | At baseline and through completion (one day)
  Time to first moderate hypoxemia and severe hypoxemia
Difference in causes of walking limitations | At baseline and through completion (one day)
  The participant is asked about factors limiting the walking distance.

CONTACTS AND LOCATIONS:
Overall Officials: Janne H Jensen, MSc, Principal Investigator — Aarhus University Hospital, Department of Physiotherapy and Occopational therapy
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bendstrup E, Hyldgaard C, Altraja A, Sjaheim T, Myllarniemi M, Gudmundsson G, Skold M, Hilberg O. Organisation of diagnosis and treatment of idiopathic pulmonary fibrosis and other interstitial lung diseases in the Nordic countries. Eur Clin Respir J. 2015 Jul 1;2. doi: 10.3402/ecrj.v2.28348. eCollection 2015. PMID 26557259
- [Background] Hansen EF, Hove JD, Bech CS, Jensen JS, Kallemose T, Vestbo J. Automated oxygen control with O2matic(R) during admission with exacerbation of COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 14;13:3997-4003. doi: 10.2147/COPD.S183762. eCollection 2018. PMID 30587955
- [Background] Hyldgaard C. A cohort study of Danish patients with interstitial lung diseases: burden, severity, treatment and survival. Dan Med J. 2015 Apr;62(4):B5069. PMID 25872544
- [Background] Jacobs SS, Krishnan JA, Lederer DJ, Ghazipura M, Hossain T, Tan AM, Carlin B, Drummond MB, Ekstrom M, Garvey C, Graney BA, Jackson B, Kallstrom T, Knight SL, Lindell K, Prieto-Centurion V, Renzoni EA, Ryerson CJ, Schneidman A, Swigris J, Upson D, Holland AE. Home Oxygen Therapy for Adults with Chronic Lung Disease. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2020 Nov 15;202(10):e121-e141. doi: 10.1164/rccm.202009-3608ST. PMID 33185464
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Background] Kofod LM, Westerdahl E, Kristensen MT, Brocki BC, Ringbaek T, Hansen EF. Effect of Automated Oxygen Titration during Walking on Dyspnea and Endurance in Chronic Hypoxemic Patients with COPD: A Randomized Crossover Trial. J Clin Med. 2021 Oct 20;10(21):4820. doi: 10.3390/jcm10214820. PMID 34768338
- [Background] Lellouche F, L'Her E, Bouchard PA, Brouillard C, Maltais F. Automatic Oxygen Titration During Walking in Subjects With COPD: A Randomized Crossover Controlled Study. Respir Care. 2016 Nov;61(11):1456-1464. doi: 10.4187/respcare.04406. Epub 2016 Oct 18. PMID 27794080
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Schneeberger T, Jarosch I, Leitl D, Gloeckl R, Hitzl W, Dennis CJ, Geyer T, Criee CP, Koczulla AR, Kenn K. Automatic oxygen titration versus constant oxygen flow rates during walking in COPD: a randomised controlled, double-blind, crossover trial. Thorax. 2023 Apr;78(4):326-334. doi: 10.1136/thoraxjnl-2020-216509. Epub 2021 Oct 16. PMID 34656996
- [Background] Vezina FA, Bouchard PA, Breton-Gagnon E, Dion G, Viglino D, Roy P, Bilodeau L, Provencher S, Denault MH, Saey D, Lellouche F, Maltais F. Automated O2 Titration Alone or With High-Flow Nasal Cannula During Walking Exercise in Chronic Lung Diseases. Respir Care. 2023 Dec 28;69(1):1-14. doi: 10.4187/respcare.10810. PMID 37491073
- [Background] Visca D, Mori L, Tsipouri V, Fleming S, Firouzi A, Bonini M, Pavitt MJ, Alfieri V, Canu S, Bonifazi M, Boccabella C, De Lauretis A, Stock CJW, Saunders P, Montgomery A, Hogben C, Stockford A, Pittet M, Brown J, Chua F, George PM, Molyneaux PL, Margaritopoulos GA, Kokosi M, Kouranos V, Russell AM, Birring SS, Chetta A, Maher TM, Cullinan P, Hopkinson NS, Banya W, Whitty JA, Adamali H, Spencer LG, Farquhar M, Sestini P, Wells AU, Renzoni EA. Effect of ambulatory oxygen on quality of life for patients with fibrotic lung disease (AmbOx): a prospective, open-label, mixed-method, crossover randomised controlled trial. Lancet Respir Med. 2018 Oct;6(10):759-770. doi: 10.1016/S2213-2600(18)30289-3. Epub 2018 Aug 28. PMID 30170904
- [Background] Vivodtzev I, L'Her E, Vottero G, Yankoff C, Tamisier R, Maltais F, Lellouche F, Pepin JL. Automated O2 titration improves exercise capacity in patients with hypercapnic chronic obstructive pulmonary disease: a randomised controlled cross-over trial. Thorax. 2019 Mar;74(3):298-301. doi: 10.1136/thoraxjnl-2018-211967. Epub 2018 Aug 30. PMID 30166425